CLINICAL TRIAL: NCT04989530
Title: Comparison of Ultrasonographic and Clinical Features of Different Energy Levels Extracorporeal Shock Wave Therapy in Plantar Fasciitis: A Randomized, Prospective, Double-blind Clinical Trial
Brief Title: Comparison of Ultrasonographic and Clinical Features of Different Energy Levels Extracorporeal Shock Wave Therapy in Plantar Fasciitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baskent University Ankara Hospital (Other)
Responsible Party: Principal Investigator, Şükran Güzel, M.D., Baskent University Ankara Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-94603339-604.01.02-46403
Record Dates: First submitted 2021-07-26; First posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Extracorporeal Shock Wave Therapy
Keywords: Extracorporeal Shock Wave Therapy; ultrasonography; plantar fasiit
MeSH Terms: interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low energy level of ESWT (Active Comparator)
  Interventions: Device: Extracorporeal Shock Wave Therapy
- medium energy level of ESWT (Active Comparator)
  Interventions: Device: Extracorporeal Shock Wave Therapy
- high energy level of ESWT (Active Comparator)
  Interventions: Device: Extracorporeal Shock Wave Therapy

INTERVENTIONS:
Device: Extracorporeal Shock Wave Therapy — different energy levels of ESWT

SUMMARY:
Plantar fasciitis is the most common cause of heel pain in adults. It received FDA approval in 2000 for ESWT in the treatment of plantar fasciitis in adults whose pain did not resolve with conservative treatment.

ESWT energy levels are categorized as high, medium and low. It is not yet clear which energy level is most effective in the clinical recovery and pain relief of plantar fasciitis after ESWT treatment. Although there are studies in the literature evaluating the effect of different energy densities in the treatment of plantar fasciitis with ESWT, there are very few studies comparing different treatment doses of ESWT.

The aim of this study was to evaluate and compare the therapeutic effects of low, medium and high energy ESWT in patients with plantar fasciitis, and also to examine the correlation between plantar fascia thickness changes ultrasonographically and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

presence of heel pain, tenderness at the insertion site of the plantar fascia on the anteromedial aspect of the calcaneal tubercle elicited by palpation, and unresponsiveness to medical treatment.

Exclusion Criteria:

history of inflammatory rheumatic disease, trauma of the foot or foot surgery, local dermatological lesion or infection, impaired peripheral circulation, a neurological disorder such as radiculopathy and neuropathy, patients with sequelae of lower extremity fracture, a congenital or acquired deformity, malignancy, cardiac pacemaker, metal implant at the application site, pregnancy, anticoagulant use for coagulopathy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Foot Function index | 1 months

SECONDARY OUTCOMES:
Plantar fasia thickness | 1 months
  Measurement of plantar fascia thickness with ultrasound

OTHER OUTCOMES:
visual analogue scale | 1 months

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University Ankara Hospital, Ankara, Turkey (Türkiye)